CLINICAL TRIAL: NCT03175575
Title: A Pilot Study to Assess How Access to a Community Garden Could Help Instigate the Adoption of Healthier Food Purchase Patterns in Deprived Neighborhood (Marseille, France)
Brief Title: Pilot Study on Community Gardens and Food Purchases in Deprived Neighborhood (Marseille, France)
Status: Completed | Type: Observational
Sponsor: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other)
Collaborators: National Research Agency, France (Other)
Responsible Party: Principal Investigator, Nicole Darmon, Senior researcher, Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement
Other Study IDs: Jassur-Marseille
Record Dates: First submitted 2017-06-01; First posted 2017-06-05 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Nutritional Quality of Food Purchases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Access to a community garden in deprived neighborhoods

SUMMARY:
The pilot study aims to investigate the place of fresh garden produce in the food supply and food practices of women in community gardens of deprived neighborhoods of Marseille, reputed to be among the poorest in the European Union. We hypothesized that access to a community garden in these neighborhoods could help instigate the adoption of healthier food patterns by gardeners and their households, and in particular, increase their consumption of fruits and vegetables.

DETAILED DESCRIPTION:
Urban community gardening was explored in terms of (i) food production, (ii) nutrition and economics, and (iii) cultural, social, and symbolic dimensions, by social and nutritional science approaches, involving informative questionnaires, semi-structured interviews, and a nutritional and economic analysis of household food supplies.

ELIGIBILITY:
Inclusion Criteria:

* Having access to a community garden in deprived neighborhoods of Marseille
* Willingness to be involved in the study
* Be in charge of the household food purchases

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Women gardeners
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2014-05-01 (Actual); Primary Completion 2014-06-30 (Actual); Study Completion 2014-06-30 (Actual)

PRIMARY OUTCOMES:
Household food supply records. | One-month
  Participants collected food purchase receipts for their household over a one-month period which constituted a detailed record of the quantities of food entering their household. They were asked to save all till receipts for foods consumed at home. To facilitate data collection, participants were given a notebook of food purchases in which they could find step-by-step instructions, example receipts, and, on the last page, an envelope in which to collect the receipts. In case of incomplete or ambiguous printed information regarding the name of the shop, the name of a food, the quantities purchased or the price paid for a food, participants were instructed to write it on the receipt. Expenditure without receipts and food items coming from the garden, or from gifts or social aid services were to be recorded in the notebook. The participants were also requested to ask other household members to keep their till receipts.

SECONDARY OUTCOMES:
Informative questionnaire | 45 min
  An informative questionnaire enabled the characterization of the 21 participants by gender, age, country of birth, number of household members, occupational status of the gardener and household members, and the gardeners' perception of their financial situation. The agronomic part of the questionnaire provided information on garden use (past gardening experience, length of time in the current plot, time working in the garden), production management (choice of crops and cultivation practices, soil knowledge and preparation, seed and plant origins, methods of crop protection, training and learning methods,exchanges with other gardeners), and garden functions as perceived by the gardeners, together with their motivations for gardening.
Comprehensive interviews | 1 hour
  To identify the unique characteristics relative to each gardener, and their aspirations and dietary practices, a comprehensive interview were conducted on 17 participants. The interviews explored three principal themes: (i) personal history and biographical elements related to gardening, (ii) links between gardening activities and food practices (food supply practices, culinary habits and skills, commensality), and (iii) social functions of the garden. Interviews were either audio-taped or recorded in writing, depending on the gardener's consent. Transcripts were analyzed and grouped thematically as prescribed by the interview guidelines. We then selected quotations based on their informative value to best illustrate the dimensions of food practices.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tharrey M, Dubois C, Maillot M, Vieux F, Mejean C, Perignon M, Darmon N. Development of the Healthy Purchase Index (HPI): a scoring system to assess the nutritional quality of household food purchases. Public Health Nutr. 2019 Apr;22(5):765-775. doi: 10.1017/S1368980018003154. Epub 2018 Nov 26. PMID 30472975